CLINICAL TRIAL: NCT01109173
Title: Clinical Evaluation of Nepafenac Ophthalmic Suspension, 0.3% for Prevention and Treatment of Ocular Inflammation and Pain After Cataract Surgery
Brief Title: Confirmatory Study Nepafenac 0.3%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-09-055
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nepafenac 0.3% (Experimental): Nepafenac Ophthalmic Suspension, 0.3%, one drop in affected eye once daily for 16 days, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery. An additional dose was administered between 30-120 minutes prior to surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.3%
- NEVANAC (Active Comparator): Nepafenac Ophthalmic Suspension, 0.1%, one drop in affected eye three times daily, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.1%
- Nepafenac Vehicle 0.3% (Placebo Comparator): Nepafenac Ophthalmic Suspension 0.3% Vehicle, one drop in affected eye once daily for 16 days, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery. An additional dose was administered between 30-120 minutes prior to surgery.
  Interventions: Other: Nepafenac Ophthalmic Suspension 0.3% Vehicle
- NEVANAC Vehicle (Placebo Comparator): Nepafenac 0.1% vehicle, one drop in affected eye three times daily, beginning one day prior to surgery, continuing on the day of surgery, and for 14 days following surgery.
  Interventions: Other: NEVANAC Vehicle

INTERVENTIONS:
Drug: Nepafenac Ophthalmic Suspension, 0.3% — Nepafenac Ophthalmic Suspension, 0.3%, one drop in affected eye once daily, for 16 days. An additional dose was administered between 30-120 minutes prior to surgery.
  Arms: Nepafenac 0.3%
Drug: Nepafenac Ophthalmic Suspension, 0.1% — Nepafenac Ophthalmic Suspension, 0.1%, one drop in affected eye three times daily, for 16 days
  Other Names: NEVANAC®
  Arms: NEVANAC
Other: Nepafenac Ophthalmic Suspension 0.3% Vehicle — Nepafenac 0.3% vehicle, one drop in affected eye once daily, for 16 days. An additional dose was administered between 30-120 minutes prior to surgery.
  Arms: Nepafenac Vehicle 0.3%
Other: NEVANAC Vehicle — Nepafenac vehicle, one drop in affected eye three times daily, for 16 days
  Arms: NEVANAC Vehicle

SUMMARY:
The purpose of this study was to assess the safety and efficacy of an investigational eye drop intended for the prevention and treatment of inflammation (swelling and redness) and pain in the eye after cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract extraction by phacoemulsification with the implantation of a posterior chamber intraocular lens;
* Patients who, in the opinion of the Investigator, would have improvement in best-corrected visual acuity after surgery;
* Able to understand and sign an informed consent;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of topical ocular, inhaled or systemic nonsteroidal anti-inflammatory drugs within 7 days of surgery, with the exception of the allowed low dose of aspirin (up to 100 mg) prior to surgery and through study exit;
* Use of topical ocular, inhaled or systemic steroids within 14 days prior to surgery and through study exit;
* History of chronic or recurrent inflammatory eye disease (eg, iritis, scleritis, uveitis, iridocyclitis, rubeosis iridis) in the operative eye;
* Diabetic retinopathy in the operative eye;
* Known or suspected allergy or hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs), or to any component of the test article;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2120 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Sager, MS, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized from 65 sites in 5 countries: US (49), Hungary (6), Italy (4), Sweden (4), and Switzerland (2).
Pre-assignment Details: Of the 2120 enrolled participants, 78 withdrew before the start of dosing. Baseline characteristics are presented on all randomized patients with at least 1 postoperative assessment (ITT): 2022.
Period: Overall Study
Arm/Group | Nepafenac 0.3% | NEVANAC | Nepafenac Vehicle 0.3% | NEVANAC Vehicle
Started | 851 | 845 | 211 | 213
Completed | 763 | 759 | 110 | 120
Not Completed | 88 | 86 | 101 | 93
Not completed — Adverse Event | 15 | 17 | 9 | 6
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Patient Decision Unrelated to Advrs Evnt | 5 | 0 | 2 | 0
Not completed — Noncompliance | 0 | 1 | 0 | 0
Not completed — Treatment Failure | 25 | 32 | 69 | 64
Not completed — Protocol Violation | 4 | 5 | 1 | 2
Not completed — Patient Did Not Use Study Medication | 34 | 26 | 11 | 7
Not completed — Not Specifiied | 5 | 4 | 9 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac 0.3% | NEVANAC | Nepafenac Vehicle 0.3% | NEVANAC Vehicle | Total
Number analyzed (Participants) | 807 | 813 | 197 | 205 | 2022
Age Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.08) | 68.8 (9.31) | 69.8 (9.31) | 68.9 (9.37) | 68.9 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 465 | 458 | 118 | 115 | 1156
  Male | 342 | 355 | 79 | 90 | 866

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Cured at Day 14
Description: Ocular inflammation was assessed by the investigator during slit lamp examination. Aqueous cells were scored on a 5-unit scale from 0 (none) to 4 (> 30 cells), and aqueous flare (protein escaping from dilated vessels) was scored on a 4-unit scale from 0 (no visible flare when compared with the normal eye) to 3 (severe - very dense flare). To be considered cured, the patient must have had a score of 0 for both cells and flare.
Time Frame: Day 14
Population: All randomized patients with at least one postoperative assessment (ITT), last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Nepafenac 0.3% | NEVANAC | Nepafenac Vehicle 0.3% | NEVANAC Vehicle
Number analyzed (Participants) | 807 | 811 | 197 | 205
percentage of participants | 68.4 | 70.0 | 34.0 | 35.6

2. Secondary Outcome: Percentage of Patients Pain-Free at Day 14
Description: Ocular pain as assessed by the investigator on a scale ranging from 0 (none) to 5 (severe). Pain-free was defined as a score of 0 on the investigator's assessment of ocular pain.
Time Frame: Day 14
Population: All randomized patients with at least one postoperative assessment (ITT), last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Nepafenac 0.3% | NEVANAC | Nepafenac Vehicle 0.3% | NEVANAC Vehicle
Number analyzed (Participants) | 807 | 811 | 197 | 205
percentage of participants | 91 | 90.9 | 49.7 | 56.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: This reporting group includes all patients who received exposure to the study medication or potential exposure to the study medication: 2042. At each study visit, the patient received an ocular exam, and any changes in ocular and systemic medications and/or systemic disease/conditions since surgery were recorded.
Arm/Group | Nepafenac 0.3% | NEVANAC | Nepafenac Vehicle 0.3% | NEVANAC Vehicle
Serious Adverse Events (participants affected / at risk) | 7/817 | 3/819 | 0/200 | 0/206
Other Adverse Events (participants affected / at risk) | 0/817 | 0/819 | 0/200 | 0/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nepafenac 0.3% (N=817) | NEVANAC (N=819) | Nepafenac Vehicle 0.3% (N=200) | NEVANAC Vehicle (N=206)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 — Not related
Brain Oedema (Nervous system disorders) | 1 | 0 | 0 | 0 — Not related
Cerebrovascular Accident (Nervous system disorders) | 1 | 1 | 0 | 0 — Not related
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — Not related
Injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 — Not related
Lung Carcinoma Cell Type Unspecified Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 — Not related
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 — Not related
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 — Not related
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 — Not related

LIMITATIONS AND CAVEATS:
This study excluded patients who were under the age of 18, had uncontrolled glaucoma, were at risk of developing macular edema (eg, diabetic retinopathy), or of childbearing potential. Therefore, results may not be generalizable to these populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.